CLINICAL TRIAL: NCT01410266
Title: The Acceptability and Feasibility of Reducing the Need for In-Clinic Follow-Up for First Trimester Medical Abortion in Moldova and Uzbekistan
Brief Title: Reducing the Need for In-Clinic Follow-Up for Medical Abortion in Moldova and Uzbekistan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6.5
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Medical Abortion, Fetus
Keywords: medical abortion; first trimester; follow-up; pregnancy test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): Standard of care includes a routine clinic visit two weeks after misoprostol administration. At the clinic visit, the woman undergoes a bimanual examination. In the event the woman fails to return for the follow-up visit, clinic procedure is followed for contacting her to determine abortion status and the need for further intervention, if any.
- Alternative follow-up (Active Comparator): At a clinic visit, before mifepristone administration, the woman completes a semi-quantitative pregnancy test. After mifepristone administration, she is provided with another pregnancy test and a checklist to be self-administered two weeks after she takes misoprostol. On an assigned date, the woman is contacted by phone by the clinic staff and asked to report on the results of both tests. The provider then confirms whether, based on the woman's responses, she should return for a follow-up visit.
  Interventions: Other: Alternative follow-up

INTERVENTIONS:
Other: Alternative follow-up — Alternative follow-up consists of a self-administered semi-quantitative pregnancy test designed to measure urine beta-hCG levels, and a self-administered questionnaire consisting of 7 questions. Results of both are reviewed by the provider to determine if in-clinic follow-up is needed.
  Other Names: semi-quantitative pregnancy test; self-administered questionnaire
  Arms: Alternative follow-up

SUMMARY:
The purpose of this study is to determine whether an alternative method of follow-up after medical abortion is acceptable and feasible for use in Moldova and Uzbekistan.

DETAILED DESCRIPTION:
Medical abortion using mifepristone and misoprostol is a highly effective procedure, but access to it may be impeded by the fact that not all women can afford or want to return for a follow-up visit. This often results in a high loss to follow-up rate. Additionally, with medical abortions of those women who do return for follow-up, higher costs are borne by both the woman and the healthcare system.

This study compares two methods of follow-up after medical abortion: standard of care versus alternative follow-up. The former involves a routine clinic visit two weeks after misoprostol administration. The latter consists of a low-sensitivity pregnancy test and a self-administered questionnaire. Based on the results of the test and questionnaire, women may be flagged as needing in-clinic follow-up or discharged from the study if their abortion is complete.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive-age woman seeking a medical abortion
* Woman in good general health
* Woman with an intrauterine pregnancy less than or equal to 63 days gestation on the day of mifepristone administration
* Woman able and willing to sign consent forms
* Woman eligible for medical abortion according to clinician's assessment
* Woman agreeing to be followed up with, by phone or at a clinic visit

Exclusion Criteria:

* Woman with a pregnancy greater than 63 days gestation on the day of mifepristone administration

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2400 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Continued, ongoing pregnancy | 1 month

SECONDARY OUTCOMES:
Percentage of women who return for follow-up | 1 month
Percentage of women receiving other treatment for ongoing pregnancy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hillary J. Bracken, PhD, MHS, MA, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (7):
- Moldova (4):
  - The Perinatalogy Center, Bălţi
  - Municipal Clinical Hospital, Chisinau
  - The National Center of Reproductive Health and Medical Genetics, Chisinau
  - The Center of Women Health "Ana", Drochia
- Uzbekistan (3):
  - Clinic #2 of Tashkent Medical Academy, Tashkent
  - Municipal Maternity House #10, Tashkent
  - Women's Wellness Center, Tashkent

REFERENCES:
- [Derived] Platais I, Tsereteli T, Comendant R, Kurbanbekova D, Winikoff B. Acceptability and feasibility of phone follow-up with a semiquantitative urine pregnancy test after medical abortion in Moldova and Uzbekistan. Contraception. 2015 Feb;91(2):178-83. doi: 10.1016/j.contraception.2014.11.004. Epub 2014 Nov 15. PMID 25497383